CLINICAL TRIAL: NCT03294460
Title: Nicotinic Receptor Genetic Variation and Alcohol Reward
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 170171; 17-AA-0171
Record Dates: First submitted 2017-09-26; First posted 2017-09-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10-09

CONDITIONS: Alcohol Drinking
Keywords: Functional Magnetic Resonance Imaging (fMRI); Alcohol Use; Polymorphism, Genetic; Magnetic Resonance Imaging (MRI); Smoking
MeSH Terms: conditions — Alcohol Drinking; Smoking | interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Alcohol self-administration (IV ethanol for sessions 1 and oral for session 2)
  Interventions: Drug: Alcohol (Oral); Drug: Alcohol (IV); Drug: Alcohol (Ethanol)

INTERVENTIONS:
Drug: Alcohol (Oral) — Oral Self-administration
Drug: Alcohol (IV) — IV Self-administration
Drug: Alcohol (Ethanol) — IV and Oral Self-administration

SUMMARY:
Background:

People with the brain disease AUD (alcohol use disorder) have a serious problem with drinking. Researchers want to study how different people react to alcohol, and how genes affect this. They will focus on a nicotine receptor gene that may increase a person s AUD risk.

Objectives:

To see if people with variations of a nicotine receptor gene take alcohol differently and have different brain responses to alcohol cues.

Eligibility:

Healthy adults ages 21 - 60. This study includes smokers and non-smokers.

Design:

Participation will be based on evaluation under the NIAAA natural history protocol (14-AA-0181) or a screening visit under this protocol.

Participants will have two 9-hour visits. They must have no alcohol or non-prescription drugs before all visits and no food or drink before the first visit.

At every visit, participants will:

* Get a light meal
* Have breath and urine tests
* Get taxi rides there and back

At visits 1, participants will:

* Have a thin plastic tube inserted in an arm and connected to a pump for alcohol infusion.
* Have sensors on their chest to monitor heart rate.
* Sit in a chair for 2.5 hours and get alcohol by pushing a button. Their breath alcohol level will be monitored.
* Answer questions about mood and effects of alcohol
* Give blood samples
* Relax at the clinic while their breath alcohol level drops

At visit 2, participants will:

* Answer questions and do computer tests
* Have an alcoholic drink and a snack
* Have a magnetic resonance imaging (MRI) scan. They will lie in a machine that takes pictures of the brain. They will do computer tasks.
* Have another drink and snack
* Relax until their alcohol level drops

Participants will have a follow-up call after each visit.

DETAILED DESCRIPTION:
Objectives:

Alcohol use disorder (AUD) is a chronic disease that has a tremendously negative impact on individuals and their families and a substantial burden on society. Research on quantitative endophenotypes such as alcohol response, and their genetic and environmental determinants, is critical to understanding the risk for AUD. There has been a great interest in examining variation in target genes that may play a mechanistic role in the expression of these endophenotypes, such the missense single-nucleotide polymorphism (SNP) in the gene encoding the 5 subunit of the nicotinic acetylcholine receptor (CHRNA5) - rs16969968. Studies have shown that CHRNA5 A-allele carriers are at greater risk for nicotine addiction and smoking-related consequences. However, little work has been done to examine the effect of this SNP on alcohol use, dependence, or alcohol response. Given the high prevalence of nicotinic receptors on dopamine (DA) neurons in brain reward regions, and the high co-use and abuse of alcohol and nicotine, these receptors may play a critical role in modulating incentive salience and reward responses to alcohol. Thus, the goal of this project is to examine the influence of CHRNA5 variation and smoking status (smokers and non-smokers) on alcohol-related phenotypes, including intravenous alcohol self-administration (IV-ASA) behavior and neuroimaging responses to cues signaling alcohol rewards.

Study Population:

This study will include 128 male and female, non-dependent drinkers, 21-60 years of age. Participants will be stratified into equally-sized groups based on their smoking status (smokers and non-smokers) and rs16969968 genotype: 1). A-allele carriers (AA or AG genotype), and 2). G-allele homozygotes (GG genotype). The study will be open to all racial and ethnic groups, as long as the individual meets the genotype criteria. Participants will be in good health as determined by medical history, physical exam, ECG, and lab tests based on evaluation under the NIAAA natural history protocol (14-AA-0181) or a screening visit under this protocol.

Design:

Participants will undergo two study procedure visits. One visit will include an IV alcohol self-administration (IV-ASA) session using the Computer-Assisted Infusion System (CAIS), which employs a physiologically-based pharmacokinetic (PBPK) model-based algorithm that allows participants free access to standardized alcohol infusions. During this session, breath alcohol concentrations (BrAC) and subjective responses will be measured as markers of the rewarding effects of alcohol. Another visit, participants will undergo a magnetic resonance imaging (MRI) session where they will be scanned while performing the Alcohol-Food Incentive Delay (AFID) task, which assesses neural processing while responding to cues signaling alcohol reward. Additional fMRI task-based scans and a resting-state scan will also be obtained.

Outcome Measures:

The following measures will be examined as a function of smoking status (smokers and non-smokers) and CHRNA5 genotype. The influence of sex, age, and recent drinking history will be examined as covariates. Primary outcome measures include: (1a) BrAC exposure (peak BrAC, number of infusions, time to binge-level BrAC) during the free-access IV-ASA; (1b) BOLD response during the AFID task in neural regions associated with alcohol reward processing, including ventral striatum, amygdala, and insula. Secondary outcome measures include; resting state functional connectivity (rsFC) between the regions associated with the salience network, including dorsal anterior cingulate cortex, insula, ventral striatum, and extended amygdala.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female participants between 21-60 years of age. [assessment: identification provided to Clinical Center Admissions office]
  2. Smoking status:

     * Smokers will have a history of at least 1 year of daily smoking, defined as individuals who smoke more than 20 uses of nicotinic products/week on average, and a cotinine level, measured by the NarcoCheck PreDosage Nicotine Test [PNT] test, of >= 2. [assessment: Smoking history questionnaire, Additional medical history, PreDosage Nicotine test]
     * Non-smokers with no history of smoking in the past year and less than 20 uses of nicotinic products lifetime.[assessment: smoking history questionnaire, Additional medical history]
  3. Inclusion criteria for women: Use of adequate method of birth control during the study, if female is sexually active and is not surgically sterilized. Adequate methods of contraception include: use of oral contraceptives; use of barrier method of contraceptive; use of an approved IUD or other long-acting reversible contraceptive [LARC]; have a male sexual partner who is surgically sterilized; or have exclusively female sexual partner[s]. Justification: To minimize the risk of administering alcohol to pregnant women, given the known effects of alcohol exposure on fetuses. [assessment: medical history]

EXCLUSION CRITERIA:

1. Current or prior history of major medical illness, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders. Justification: Many illnesses may alter the neuropsychological effects of alcohol as well as MRI measures. [assessment: clinically significant findings on medical history and physical exam, ECG, laboratory tests]
2. Positive hepatitis [A, B antigen, or C], or HIV test at screening. Justification: Hepatitis can alter liver function and alcohol pharmacokinetics. HIV infection can alter brain function. [assessment: laboratory tests]
3. Current [past 12 months] history of psychiatric disorders, including depressive disorder, bipolar disorder, or anxiety disorders. Justification: Concurrent psychopathology can alter brain function and alcohol response. [assessment: SCID interview]
4. Lifetime history of psychotic disorders, obsessive compulsive disorder [OCD], post-traumatic stress disorder [PTSD], or eating disorder. Justification: These disorders can have long-term effects on brain function and alcohol response. [assessment: SCID interview]
5. Current or lifetime diagnosis of alcohol or substance use disorder. Past mild AUD or past mild SUD with no current symptoms for atleast 2 years will not be exclusionary. Justification: History of moderate to severe alcohol or substance use disorder will impact brain function and alcohol response. We do not anticipate past mild AUD or SUD in remission for 2+ years would have such impact on brain function and alcohol response. We will examine this in our exploratory analysis. We will also do a follow-up telephone/teleheath visit with these participants to assess any changes in alcohol or substance use or problems related to their participantion in the study [assessment: SCID interview]
6. Currently seeking treatment for alcohol use disorders. Justification: It would be unethical to administer alcohol to individuals seeking treatment for alcohol problems. Also, this study does not provide treatment for individuals with alcohol use disorder. [assessment: medical history]
7. History of significant withdrawal symptoms or presence of clinically significant withdrawal symptoms [Clinical Institute Withdrawal Assessment [CIWA] score > 8] at screening. Justification: Withdrawal symptoms would be indicative of alcohol use disorder, which is already an exclusion criteria. Additionally, withdrawal symptoms would be a major safety concern for participants, and a major confound in the assessment of alcohol response and brain function. [assessment: CIWA assessment]
8. Non-drinkers [alcohol-naive individuals or current abstainers] or individuals with no experience drinking 5 or more drinks on one occasion in their lifetime. Justification: It would be unethical to administer alcohol to individuals that do not drink alcohol. [assessment: Timeline Follow Back, Lifetime Drinking History, Additional History Form and medical history]
9. Positive result on urine drug screen or positive breathalyzer during screening visit. Positive urine drug screen or breathalyzer reading during more than 1 study visit will result in participant withdrawal from the study. Justification: Current or recent exposure to alcohol or drugs of abuse could impact brain function and alcohol response. [assessment: laboratory tests and breathalyzer test.
10. Current or prior history of alcohol-induced flushing reactions, including rapid reddening of the face, rapid heart rate and breathing, and nausea after 1 or 2 drinks. Justification: It would not be safe to administer alcohol to individuals with the highly aversive flushing response to alcohol. [assessment: alcohol flushing questionnaire]
11. Medication exclusion criteria:

    * Use of prescription or OTC medications known to interact with alcohol 2 weeks prior to screening or screening update visit. These include, but may not be limited to: isosorbide; nitroglycerine; benzodiazepines; warfarin; anti-depressants such as amitriptyline, clomipramine and nefazodone; anti-diabetes medications such as glyburide, metformin and tolbutamide; H2-antagonists for heartburn such as famotidine, cimetidine and ranitidine; muscle relaxants; anti-epileptics including phenytoin and phenobarbital; codeine and opioid analgesics including Darvocet, Percocet and hydrocodone;
    * regular (more than once a week) or prescribed use of the following medications and unable to refrain from these medications for 48 hours prior to study visits: anti-histamines, pain medicines, and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib, and naproxen.
    * Use of medications known to inhibit or induce enzymes that metabolize alcohol for 4 weeks prior to screening. These include chlorzoxazone, isoniazid, metronidazole, and disulfiram.
    * Use of drugs known to affect hemodynamic response 2 weeks prior to screening or screening update visit. These include antihypertensives, insulin, and thyroid medications.

    Note that any discontinuation of medications will only be done at the recommendation of a physician. [assessment: medical history and physical exam]
12. Exclusion criteria for MRI:

    * Left-handedness [Edinburgh Handedness Scale]. Justification: To avoid lateralized effects on brain function measures and reduce potential variance in MRI signals.
    * Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head [including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments].
    * Fear of enclosed spaces. Justification: To minimize risk and discomfort.
    * Inability to lie comfortable on back for up to 2 hours in the MRI scanner. Justification: To minimize risk and discomfort. [assessment: NIAAA MRI Safety Screening Questionnaire]
13. Exclusion criteria for women: Justification: To minimize the risk of administering alcohol to pregnant or nursing women, given the known effects of alcohol exposure on fetuses and infants.

    * Pregnant [assessment: urine beta-hCG test at screening]. Women must also test negative on urine beta-hCG test at the start of every study visit.
    * Breast-feeding [assessment: medical history and physical exam].

Screen Failures:

Screen failures are defined as participants who consent to participate in the clinical trial but are not subsequently assigned to the study intervention or entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants, to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse event (SAE).

Individuals who do not meet the criteria for participation in this trial (screen failure) because of a positive drug test, positive pregnancy test or positive breathalyzer reading may be rescreened. Rescreened participants should be assigned the same participant number as for the initial screening.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of CHRNA5 (rs16969968) genetic variation on neural correlates of incentive salience for alcohol, as measured by BOLD response during the Alcohol-Food Incentive Delay (AFID) task using fMRI. | 3 hours
  The following measures will be examined as a function of smoking status (smokers and non-smokers) and CHRNA5 genotype. The influence of sex, age, and recent drinking history will be examined as covariates. Primary outcome measures include: (1a) BrAC exposure (peak BrAC, number of infusions, time to binge-level BrAC) during the free-access IV-ASA; (1b) BOLD response during the AFID task in neural regions associated with alcohol reward processing, including ventral striatum, amygdala, and insula. Secondary outcome measures include: (2a) resting state functional connectivity (rsFC) between the regions associated with the salience network, including dorsal anterior cingulate cortex, ventral striatum, and extended amygdala; (2b) preferred rate of self-infusion during the second IV-ASA session.
To examine the effect of CHRNA5 (rs16969968) genetic variation on IV alcohol self-administration, as measured by BrAC exposure (peak BrAC, number of infusions, time to binge-level) in non-smoking, non-dependent drinkers. | 3 hours
  The following measures will be examined as a function of smoking status (smokers and non-smokers) and CHRNA5 genotype. The influence of sex, age, and recent drinking history will be examined as covariates. Primary outcome measures include: (1a) BrAC exposure (peak BrAC, number of infusions, time to binge-level BrAC) during the free-access IV-ASA; (1b) BOLD response during the AFID task in neural regions associated with alcohol reward processing, including ventral striatum, amygdala, and insula. Secondary outcome measures include: (2a) resting state functional connectivity (rsFC) between the regions associated with the salience network, including dorsal anterior cingulate cortex, ventral striatum, and extended amygdala; (2b) preferred rate of self-infusion during the second IV-ASA session.

SECONDARY OUTCOMES:
To examine the relationship between fMRI measures (BOLD response during AFID and rsFC measures) and IV alcohol self-administration, and any differences in the degree of association among these measures by CHRNA5 genotype. | 3 hours
To examine the effect of CHRNA5 (rs16969968) genetic variation on the rate of IV alcohol self-administration, as measured by the preferred rate during the second IV-ASA session in non-smoking, non-dependent drinkers. | 3 hours
To examine the effect of CHRNA5 (rs16969968) genetic variation on resting-state functional connectivity (rsFC) among brain regions associated with the salience network, including dorsal anterior cingulate cortex, ventral striatum and extended am... | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-AA-0171.html